CLINICAL TRIAL: NCT04449744
Title: Effects of Remote Motivational Enhancement & MySafeRx on Post-Detox Engagement and Retention in Buprenorphine Treatment (MySafeRx) - A Pilot Study
Brief Title: Evaluating Adaptive Dispenser Initiation Protocols for MySafeRx During Post-detox Buprenorphine Treatment- a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Cambridge Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00038163 - Pilot; R01CE003039 (NIH)
Record Dates: First submitted 2020-06-11; First posted 2020-06-29 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2020-05

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MySafeRx Group A-(coaching + medication dispenser) (Active Comparator): The MySafeRx™ platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of buprenorphine/naloxone medication within a secure electronic pill dispenser, and a standardized protocol for supervising self-administration of medication via videoconferencing.
  Interventions: Other: MySafeRx Inspire Plus
- MySafeRx Group B-(coaching + dispenser based on clinical need) (Experimental): The MySafeRx™ platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of buprenorphine/naloxone medication within a manual lockbox, and a standardized protocol for supervising self-administration of medication via videoconferencing. Participants will be assessed bi-weekly by their clinical team for substance abuse, coaching and medication adherence, compliance with urine drug screen policies, safety/ risk or mental health concerns, and diversion. Based on clinical need, the participant may be assigned an electronic pill dispenser for the duration of the study.
  Interventions: Other: MySafeRx Inspire Flex

INTERVENTIONS:
Other: MySafeRx Inspire Plus — The MySafeRx™ platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of buprenorphine/naloxone medication within a secure electronic pill dispenser, and a standardized protocol for supervising self-administration of medication via videoconferencing.
  Arms: MySafeRx Group A-(coaching + medication dispenser)
Other: MySafeRx Inspire Flex — The MySafeRx™ platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of buprenorphine/naloxone medication within a secure electronic pill dispenser, and a standardized protocol for supervising self-administration of medication via videoconferencing. Based on clinical need, the participant may be assigned an electronic pill dispenser for the duration of the study by their clinical team.
  Arms: MySafeRx Group B-(coaching + dispenser based on clinical need)

SUMMARY:
Opioid overdoses are a significant problem nationwide and novel interventions that can prevent overdose by improving buprenorphine treatment for opioid use disorder are a public health priority. This study will both investigate the effects of starting remote motivational enhancement during inpatient detoxification on rates of engagement in Buprenorphine/ Naloxone (B/N) treatment and evaluate the impact of MySafeRx, a mobile device application which integrates remote motivational coaching with daily observed dosing from secure electronic pill dispensers at home via videoconference, on treatment retention and overdose prevention. Broad dissemination of this new intervention could help communities across the nation expand and advance their capacity to increase B/N treatment engagement and retention, enhance medication adherence, and prevent overdose.

DETAILED DESCRIPTION:
The objective of this study is to evaluate an innovative strategy among opioid use disorder patients being discharged from detox. This study will evaluate the extent to which remote motivational enhancement sessions via videoconference and the option for flexible daily dosing at home with MySafeRx can improve engagement and retention with Buprenorphine/Naloxone (B/N) treatment after detox in a county where access to B/N treatment has primarily been provided with in-person, onsite, daily dosing. This study seeks to expand the investigators understanding about what works to prevent opioid overdose by evaluating the effects of remote motivational enhancement (RME) sessions provided via videoconferencing at an inpatient detox facility and during early treatment in order to increase treatment engagement with daily outpatient supervised-dosing of B/N. Participants will use an Android smartphone device to access the MySafeRx app and complete their daily motivational interview sessions. In addition, the study seeks to evaluate the effects of using a locked medication dispenser. The role of the dispenser has not been fully evaluated in the past, and evaluation is needed to determine if the dispenser is necessary at the start of a treatment program or only in response to those participants having issues with adherence or participants that are struggling. This pilot study will generate new knowledge about the most effective way to prevent overdose and engage patients in B/N treatment with observed daily dosing.

Hypothesis:

The investigators will examine whether acceptable levels of satisfaction with the MySafeRx platform, specifically the electronic pill dispenser, are achieved at the end of the pilot period.

Primary Aim:

Aim 1: To assess the acceptability of the electronic medication dispenser and evaluate the impact of using an alternative adaptive assessment-based procedure, by comparing MySafeRx Group A (all participants in MySafeRx receive an electronic pill dispenser at the start) and MySafeRx Group B (participants only receive the electronic medication dispensers based on clinical evaluation and need after assessment at regular time intervals).

Secondary Aims:

Aim 2: To examine the differences in positive urine toxicology screens between MySafeRx Group A (coaching + medication dispenser) and MySafeRx Group B (coaching + medication dispenser based on clinical need)

Aim 3: To examine medication adherence to B/N by assessing the differences between MySafeRx Group A (coaching + medication dispenser) and MySafeRx Group B (coaching + medication dispenser based on clinical need) in the total number of observed B/N doses taken in the first 28 days, between weeks 3-6.

Aim 4: To examine the differential impact of two tele-health interventions of MySafeRx Group A (coaching + medication dispenser) and MySafeRx Group B (coaching + medication dispenser based on clinical need) on retention in outpatient buprenorphine treatment with B/N dosing through 24 weeks.

Exploratory COVID-19 Objectives:

Aim 5: To examine the differences of COVID-19 infection between MySafeRx Group A and MySafeRx Group B and compare with ACTS overall program incidence rate during the time period.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* opioid use disorder
* stepping down from inpatient detox services
* willing to engage in daily outpatient supervised dosing of B/N.

Exclusion Criteria:

* cognitively impaired (Unable to complete consent quiz at 90% accuracy AND MOCA < 25/30 relative exclusion requiring PI approval, absolute exclusion for MOCA<21/30)
* homeless
* reporting active homicidal or suicidal ideation with an imminent plan
* current mania or psychosis
* expected incarceration in next 3 months (those that are incarcerated during the study will be removed from the study)
* unable or unwilling to use a mobile device
* medical contraindication to BUP
* unable to complete baseline assessments
* unstable medical illness who expect hospitalization in the next 3 months pregnant women (if a patient becomes pregnant while participating in this study, they will be withdrawn)
* prisoners
* court-ordered individuals
* unable to speak or read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of Medication Dispenser | 12 weeks
  To examine the acceptability of the electronic medication dispenser and evaluate the impact of using an alternative adaptive assessment-based procedure, by comparing. MySafeRx Group A (all participants in MySafeRx receive an electronic pill dispenser at the start) and MySafeRx Group B (participants only receive the electronic medication dispensers based on clinical evaluation and need after assessment at regular time intervals). MySafeRx Participant Satisfaction Survey to assess for acceptability of electronic dispenser.

SECONDARY OUTCOMES:
Biochemically-Confirmed Illicit Opioid Use | 24 weeks
  To examine the differences in illicit opioid use throughout the 24 weeks of the study as measured by urine toxicology testing every 4 weeks between MySafeRx Group A (coaching + medication dispenser) and MySafeRx Group B (coaching + medication dispenser based on clinical need). Positive results for fentanyl, opiates, methadone and oxycodone will be measured at 6 time points every 4 weeks.
Outpatient Buprenorphine Medication Adherence | 12 weeks
  To examine medication adherence to Buprenorphine (B/N) by assessing the differences between MySafeRx Group A (coaching + medication dispenser) and MySafeRx Group B (coaching + medication dispenser based on clinical need) in the total number of observed B/N doses taken in the first 12 weeks. To be measured by examining adherence data from the study site EHR system and MySafeRx application.
Outpatient Buprenorphine Treatment Engagement/ Retention | 24 weeks
  To examine the differential impact of two tele-health interventions of MySafeRx Group A (coaching + medication dispenser) and MySafeRx Group B (coaching + medication dispenser based on clinical need) on retention in outpatient buprenorphine treatment with B/N dosing through 24 weeks.To be measured by examining adherence data from the study site EHR system.

OTHER OUTCOMES:
Proportion of days engaged in observed daily dosing of Buprenorphine during first 2 weeks. | Between the day after detox discharge to two-week time point
  To examine the difference in engagement defined as the proportion of participants assigned to Group A or Group B, who have an observed B/N dosing on at least 10 out of the first 14 days.
COVID-19 Infections | 24 weeks
  To examine the differences of COVID-19 infection between MySafeRx Group A (coaching + medication dispenser) MySafeRx Group B in comparison with the local treatment sites overall program incidence rate during the time period. Measured with COVID-19 self-report survey.
Number of Opioid Overdoses (Total of non-fatal self-report, clinic-reported, and fatal) | 24 weeks
  To examine the effect of RME + MySafeRx Group A (coaching + medication dispenser) + MySafeRx Group B (coaching + medication dispenser based on clinical need) on the number of self-reported, county coroner reported, and clinic-reported opioid overdoses, throughout the 24 weeks of the study.
Opioid-Related Death Rates | 24 weeks
  To examine the effect of RME + MySafeRx Group A (coaching + medication dispenser) + MySafeRx Group B (coaching + medication dispenser based on clinical need) on all opioid-related deaths (in which opioids were present at time of death), as collected through county coroner reports and community network reports, throughout the 24 weeks of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, PhD, Principal Investigator — University of South Florida; Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- ACTS Adult Addiction Receiving Facility (AARF), Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data related to our outcome measures will be included in the IPD sharing plan, in addition to our study protocol, informed consent, and analytic plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication and within 12 months of completion of the analysis of study primary aims, anonymous and de-identified data will be made available at the Open Science Framework (http://osf.io/) and/or Harvard Dataverse (https://dataverse.harvard.edu/) so that other investigators can verify or follow-up on the reported analyses.
Access Criteria: Anonymous and de-identified data will be stored on the Open Science Framework website (http://osf.io/) and/or Harvard Dataverse to be made available to other researchers to verify the research results. Before publication, only USF and CHA investigators will have direct access to the data, and only the CHA HERLab investigators will have access to the analyses.

REFERENCES:
- [Background] Schuman-Olivier Z, Borodovsky JT, Steinkamp J, Munir Q, Butler K, Greene MA, Goldblatt J, Xie HY, Marsch LA. MySafeRx: a mobile technology platform integrating motivational coaching, adherence monitoring, and electronic pill dispensing for enhancing buprenorphine/naloxone adherence during opioid use disorder treatment: a pilot study. Addict Sci Clin Pract. 2018 Sep 24;13(1):21. doi: 10.1186/s13722-018-0122-4. PMID 30249279

DOCUMENTS (1):
  • Informed Consent Form (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT04449744/ICF_000.pdf